CLINICAL TRIAL: NCT01609829
Title: iCOMtrain, Development and Evaluation of a Combined Training of Technical and Non-Technical Skills During the Management of Simulated Incidents in Intensive Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: iCOMtrain
Record Dates: First submitted 2012-05-29; First posted 2012-06-01 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Technical and Non-technical Training of Airway Management on ICU

STUDY DESIGN:
Observational Model: Cohort

INTERVENTIONS:
Procedure: SAFE (situation, all together, fly on, evaluate) — Video-assisted, structured debriefing after simulated critical airway-events.

SUMMARY:
The normal, the anticipated difficult and the unanticipated difficult airway are trained in the patient safety simulation center (University Hospital Zürich) and the training is being observed by video installation.

Step 1: normal airway (Phantom), technical training

Step 2: difficult airway (SimMan 3G), technical training

Step 3: Simulation of normal and difficult airway management on ICU (SimMan 3G), technical and non-technical (CRM - crew resource management) training.

ELIGIBILITY:
Inclusion criteria:

* doctors and nurses with a minimum of 12 moths of work experience.

Exclusion criteria:

* staff members that deny participation or don't meet the inclusion criteria

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Doctors and nurses working on the surcical ICU.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bastian Grande, MD, Principal Investigator — University Childrens Hospital Zurich, Anesthesiology
Locations (1):
- University Children's Hospital, Anesthesiology, Zurich, Canton of Zurich, Switzerland